CLINICAL TRIAL: NCT02154087
Title: A Phase 2 Exploratory Pharmacodynamic Study of HP802-247 in Venous Leg Ulcers
Acronym: MOA 034
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: based on outcome of previous study
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 802-247-09-034
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Venous Leg Ulcers
Keywords: Venous leg ulcer; Ulcer; Venous stasis; Compression
MeSH Terms: conditions — Varicose Ulcer; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HP802-247 (Experimental)
  Interventions: Biological: HP802-247

INTERVENTIONS:
Biological: HP802-247 — 260 µL (130 µL, one spray, of each component) containing 0.5 x 10.6 cells per mL, alternating weekly with Vehicle

SUMMARY:
Assess the influence of HP802-247 on biochemical and cellular markers of inflammation in chronic venous leg ulcers

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Age ≥ 18 years and of either sex
* Willing to comply with protocol instructions, including allowing all study assessments
* Have a venous leg ulcer (VLU) between the knee and ankle (at or above the malleolus), with a surface area ≥ 4.0 cm x cm and ≤ 15.0 cm x cm
* Venous insufficiency confirmed by duplex Doppler ultrasound examination for valvular or venous incompetence
* Arterial supply adequacy confirmed
* Target ulcer involves a full thickness skin loss, but WITHOUT exposure of tendon, muscle, or bone
* Target ulcer duration ≥ 12 weeks but ≤ 104 weeks (24 months).
* Acceptable state of health and nutrition

Exclusion Criteria:

* History of anaphylaxis, serum sickness, or erythema multiforme reaction to aprotinin, bovine serum albumin or bovine serum proteins, penicillin, streptomycin, amphotericin B or any other component of HP802-247,or known sensitivity to Iodine
* Prior diagnosis of Systemic Lupus Erythematosus with elevated anti-DNA antibody titers, Buerger's disease (thromboangiitis obliterans), current diagnosis of vasculitis, or current diagnosis of claudication
* Therapy with another investigational agent within thirty (30) days of Screening, or during the study, or any participation in a previous HP802-247 trial
* A target ulcer of non-venous etiologies (e.g., sickle cell anemia, necrobiosis lipoidica diabeticorum, pyoderma gangrenosum, vasculopathic or vasculitic)
* Documented history of osteomyelitis at the target wound location within 6 months preceding the Screening Visit
* Refusal of or inability to tolerate compression therapy
* Therapy of the target ulcer with Collagenase Santyl® ointment, autologous skin graft, biological dressings or living cell products (e.g., Oasis®, Apligraf™, Dermagraft™) within 30 days preceding the Screening Visit
* Therapy of the target ulcer with topical growth factors within 1 week preceding the Screening Visit
* Current therapy with systemic antibiotics
* Current systemic therapy with cytotoxic drugs
* Current therapy with chronic (> 10 days) oral corticosteroids
* Current therapy with TNFα inhibitors
* History of cancer in the preceding 5 years (other than carcinoma in situ of the cervix or adequately treated non-melanoma skin cancers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Smith & Nephew Biotherapeutics; Chief Medical Officer
Locations (1):
- Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a single US investigation site, between July 14,2014 and November 2, 2014.
Pre-assignment Details: Subjects entered a 2-week run-in; subjects whose wound radius decreased by < 0.349 cm/2weeks and met all other inclusion/exclusion (I/E) criteria were eligible for randomization.
  HP802-247
Groups:
- HP802-247: HP802-247: 260 µL (130 µL, one spray, of each component) containing 0.5 x 10.6 cells per mL, alternating weekly with Vehicle
  HP802-247 (fibrinogen solution & thrombin solution containing living, irradiated, growth-arrested keratinocytes and fibroblasts) applied every 2 weeks, with Vehicle (fibrinogen solution & acellular thrombin solution) on alternate weeks, for up to 12 weeks, or until wound closure occurred, which ever came first
Period: Overall Study
Arm/Group | HP802-247
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Termination | 1

BASELINE CHARACTERISTICS:
Arm/Group | HP802-247
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Determine Change From Baseline in Cell Numbers in Subjects With VLU Following the First Dose of HP802-247
Description: The following mediators were to be measured for the chronic ulcer stage: IL-1β, IL-6, TNF-α, IFN, MMP-2, and MMP-9, and the following for the resolving ulcer stage: PGE-2, Lipoxin, GM-CSF, TGFβ, IL-10, LL-37, Indoleamine 2,3-Dioxygenase (IDO), and Arginase (ARG-1). Each of the soluble mediators were to be plotted versus measurement time point [i.e., (pre-study run-in visit (RV)1), baseline (RV3), study visit (SV)2, and SV3]) and by subjects' quartile of percent reduction (%) in target wound area at SV3 from baseline (RV3).
Time Frame: Wound fluid samples were to be collected one week after the initial dose of HP802-247.
Population: Due to the failure of HP802-247-09-029 to show superiority over its vehicle in study 802-247-09-029, this study was terminated after enrollment of one of the proposed 25 subjects. No data was collected.
Arm/Group | HP802-247
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events were not monitored for the participants due to the early termination of the study.
Arm/Group | HP802-247
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less